CLINICAL TRIAL: NCT05862701
Title: Comparison of Topical 5% Permethrin and Topical 10% Sulfur in the Treatment of Scabies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Dr Aleena Nasir, Principal Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMH Abbottabad Dermatology
Record Dates: First submitted 2023-03-28; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Scabies
Keywords: scabies; permethrin; ointment; therapeutics
MeSH Terms: conditions — Scabies | interventions — Permethrin; Sulfur

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Permethrin (Active Comparator): Group A treated with application of topical 5% permethrin cream twice with one week interval. Follow-up at 1, 2 and 4 weeks
  Interventions: Drug: Permethrin
- Sulfur (Active Comparator): Group B treated with 10% sulfur ointment for two or three weeks. Follow-up at 1, 2 and 4 weeks
  Interventions: Drug: Sulphur

INTERVENTIONS:
Drug: Permethrin — 5% permethrin cream
  Other Names: Lotrix
  Arms: Permethrin
Drug: Sulphur — 10% Sulfur ointment
  Other Names: Scabion
  Arms: Sulfur

SUMMARY:
Sarcoptes scabiei is responsible for a skin infection called scabies. Permethrin is most widely used anti-scabicidel drug and is taken as drug of choice because of its efficacy, safety and patient's compliance. Sulfur 6-33%, as cream, ointment or lotion, is recommended by the European guidelines as an effective alternative treatment and is among the oldest treatments used for scabies. It is recommended to be applied for 3 consecutive days.

Both permethrin and sulfur have been shown in previous studies to be superior to other anti-scabietic drugs in terms of efficacy. Two studies showed that permethrin was more efficacious than sulfur, whereas a single study showed otherwise. Therefore, only a few studies are available to find a direct comparison of the efficacy of topical 5% permethrin and topical 10% sulfur in the treatment of scabies and none of them have been carried out in Pakistan. The objective of the study is to compare the efficacy of topical 5% permethrin cream and sulfur 10% ointment in the treatment of scabies.

DETAILED DESCRIPTION:
The mite named as Sarcoptes scabiei is responsible for a skin infection called scabies. This parasite is a tiny mite that is commonly not visible without a microscope and is present at stratum corneum level in the skin. It burrows in the patient's skin and causes this contagious infection.

Permethrin is an insecticide that kills the mites and permethrin 5% cream is among the commonly used drugs for scabies. It is most widely used and taken as drug of choice because of its efficacy, safety and patient's compliance. European guidelines for the management of scabies recommend 5% permethrin cream to be applied from head to toe for 8-12 hours before washing it off and treatment to be repeated after 7 to 14 days. Sulfur 6-33%, as cream, ointment or lotion, is recommended by the European guidelines as an effective alternative treatment and is among the oldest treatments used for scabies. It is recommended to be applied for 3 consecutive days. Topical Sulfur 5-10% ointment (precipitated sulfur) is among the safe and cost effective treatment options for scabies. The toxicity of sulfur ointment is low and therefore can be used in pregnancy and in children. Efficacy ratio although not very clear from previous data now shows that it cures scabies especially the type called Norwegian scabies. It is recommended to be applied on whole body for 3 successive days.

A lot of therapeutic options have been used to treat scabies but still there is a need to study those drugs for their efficacy and duration of treatment to eradicate the scabies completely from the patients and their environment. In a study done in 1994, when the use of permethrin was not very common, there were reports of killing the mites within one hour in vitro but in year 2000, it was reported that 35% mites were still alive even after 3 hours. Both permethrin and sulfur have been shown in previous studies to be superior to other anti-scabietic drugs in terms of efficacy. Two studies showed that permethrin was more efficacious than sulfur, whereas a single study showed otherwise.

Therefore, only a few studies are available to find a direct comparison of the efficacy of topical 5% permethrin and topical 10% sulfur in the treatment of scabies and none of them have been carried out in Pakistan. The objective of the study was to compare the efficacy of topical 5% permethrin cream and sulfur 10% ointment in the treatment of scabies. The hypothesis of the study was that there is a significant difference in efficacies of 5% permethrin cream and 10% sulfur ointment in the treatment of scabies. The study will help the dermatologists to develop better drug treatment strategies for their patients, and will also assist in curbing the spread of this disease to the community hence reducing its burden.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* diagnosis with scabies mites

Exclusion Criteria:

* history of allergy to any drug
* pregnancy
* lactation
* history of severe systemic disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Symptomatic Impovement | 4 weeks
  Efficacy was assessed by clinical improvement of previous lesionss assessed by visual analogue scale
No new lesions formation | 4 weeks
  Efficacy was assessed by absence of new skin lesions assessed by visual analogue scale
Absence of Pruritus | 4 weeks
  Efficacy was assessed by absence of Pruritus assessed by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Abbottabad, Abbottābād, Khyber Pakhtunkhawa, Pakistan